CLINICAL TRIAL: NCT01456884
Title: Music Therapy as a Pain Modifying Intervention in Children With Life-limiting Neurological Impairments and Metabolic Conditions
Brief Title: Music Therapy for Pain Modification in Pediatric Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: American Music Therapy Association (Other); Canuck Place Children's Hospice (Unknown); Child and Family Research Institute (Other); BC Women's Hospital and Health Centre (Unknown)
Responsible Party: Principal Investigator, Liisa Holsti, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H11-02440
Record Dates: First submitted 2011-09-29; First posted 2011-10-21 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Neurological Impairment
Keywords: Music therapy; Infants; Children; Adolescents; pediatric; palliative care; neurological impairment; metabolic condition; pain management
MeSH Terms: conditions — Neurologic Manifestations; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Live - Vibroacoustic (Experimental): Treatment order A: live guitar and vocal music therapy on day one, vibroacoustic music therapy on day two.
  Interventions: Behavioral: Live guitar and vocal music therapy; Behavioral: Vibroacoustic Music Therapy
- Vibroacoustic - Live (Experimental): Treatment order B: vibroacoustic music therapy live guitar on day one, and vocal music therapy on day two.
  Interventions: Behavioral: Live guitar and vocal music therapy; Behavioral: Vibroacoustic Music Therapy

INTERVENTIONS:
Behavioral: Live guitar and vocal music therapy — Live guitar and vocal music therapy. Subject is passive recipient for 30 minutes.
Behavioral: Vibroacoustic Music Therapy — 30 minutes using vibroacoustic mat.
  Other Names: Somatron

SUMMARY:
The purpose of this within-subjects randomized controlled trial is to determine whether two music therapy interventions are efficacious in reducing pain symptoms, in order to improve the quality of care for children in pediatric hospice. The investigators hypothesize that both music therapy interventions, live guitar and vocal intervention and vibroacoustic intervention, will reduce behavioural pain scores and that behavioural pain scores will correlate with physiological outcome measures.

DETAILED DESCRIPTION:
Effective pain management in pediatric palliative care is a quality of life issue for patients, families and professionals. Current research supports the use of music therapy to assist with pain management in pediatric medical settings. However, little research has been done to explore the use of music therapy for reducing pain in children with life-limiting neurological impairments or metabolic conditions.

As the first known project to examine the effects of music therapy on pain symptoms with children who have life-limiting neurological impairments or metabolic disorders, this study will expand the evidence-base for practice with this population. It is imperative that an evidence base for music therapy in this area be established, so that the most effective interventions can be provided to these vulnerable children.

ELIGIBILITY:
Inclusion Criteria:

* Children, ages 1-19, who have been diagnosed with life-limiting neurological impairments and metabolic conditions
* Cognitive functioning level of one year or less will be enrolled in the study
* Receiving respite or symptom management care at the time of admission to the Canuck Place Children's Hospice
* Guardians must be able to provide written consent in English; interpreters will be available if a guardian needs clarification on specific points.

Exclusion Criteria:

* Children who are actively dying (i.e. admitted for end-of-life care or determined by physicians to require immediate end-of-life care)
* Any history of adverse responses to live or recorded music or to vibroacoustic stimulation
* Severe to profound hearing impairment will be excluded.

Ages: 12 Months to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2012-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Behavioural Pain Scores | Participants will be observed for a total of 3 hours during one hospice admission, an expected average of one week
  Non-communicating children's pain checklist scores.

SECONDARY OUTCOMES:
Physiological measures | Participants will be observed for a total of 3 hours during one hospice admission, an expected average of one week
  Heart rate, oxygen saturation, skin conductance

CONTACTS AND LOCATIONS:
Overall Officials: Liisa Holsti, PhD, Principal Investigator — University of British Columbia; Beth Clark, MM, Study Director — Canuck Place Children's Hospice; Harold Siden, MD, Study Director — Canuck Place Children's Hospice
Locations (1):
- Canuck Place Children's Hospice, Vancouver, British Columbia, Canada